CLINICAL TRIAL: NCT02286076
Title: Impact of Laparoscopic Endometrioma Stripping Surgery on Fertility: Pre- Operative and Post- Operative Changes of Serum Anti-mullerian Hormone Levels
Brief Title: Influence of Laparoscopic Endometrioma Stripping Surgery on Serum Anti-mullerian Hormone Levels
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Svetlana Spremovic- Radjenovic, Professor of Gynecology and Obstetrics, Clinical Centre of Serbia
Other Study IDs: 1040/30
Record Dates: First submitted 2014-11-01; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Endometriosis
Keywords: endometrioma; laparoscopy; ovarian reserve
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The endometrioma specimens that will be obtained from operation will be submitted for pathology examination
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare changes in follicular ovarian reserve in women before and six months after laparoscopic operation: endometrioma stripping surgery. Also, to compare follicular ovarian reserve in women with endometrioma(s) with follicular ovarian reserve of healthy infertile women of the same age group.

DETAILED DESCRIPTION:
In order to investigate the impact of laparoscopic stripping surgery on follicular ovarian reserve, blood samples will be obtained before the operation, from 2nd to 5th day of the menstrual cycle, to determine levels of endocrine markers of ovarian reserve (FSH, E2, AMH and Inhibin B). Cancer antigen 125 (CA -125) and IL-6 will be measured also. US markers (antral follicular count- AFC) will be obtained at the same time as endocrine markers. All laparoscopic stripping surgery will be performed during the early or middle follicular phases of menstrual cycle, under general anesthesia, by the same team of gynecological endoscopist. The cyst wall will be completely stripped off from the normal ovarian tissue by traction and opposite traction with two grasping forceps. Hemostasis will be achieved using bipolar forceps electrocoagulation. All endometrioma specimens that will be obtained from operation will be submitted for pathology examination. One and six months after the laparoscopic cystectomy, from 2nd to 5th day of menstrual cycle, we will determine endocrine markers of ovarian reserve and levels of CA 125 and IL-6.

The control group will be consisted of healthy women with infertility problem. From the second to the fifth day of the menstrual cycle we will take blood samples to determinate endocrine markers of follicular ovarian reserve: AMH, FSH, E2, Inhibin B.

ELIGIBILITY:
Inclusion Criteria:Study group: Women with endometrioma(s)

* Age: 18- 42 years of age
* Regular menstrual cycles defined as cycle length between 25- 35 days
* Ultrasound made diagnosis of endometrioma unilateral or bilateral ≥4 cm in diameter.
* Laparoscopically and histologically confirmed diagnosis.
* Agreement to be enrolled in the study

Control group: Healthy reproductive aged women with tubal, unexplained or male infertility.

-

Exclusion Criteria:

* Previous ovarian surgery
* Suspicious of malignancy
* Known endocrine disorder or other chronic diseases.
* Use of oral contraceptive drug, gonadotropin- releasing hormone (GnRH) agonist/ antagonist, or other drugs related with ovarian function in at least 3 months before surgery.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: study group: patients with diagnosed endometrioma(s) in one ovary or in both ovaries, in reproductive years, otherwise healthy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of follicle-stimulating hormone (FSH) | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the endocrine marker of ovarian reserve
Change of estradiol (E2) levels | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the endocrine marker of ovarian reserve
Change of Anti-mullerian hormone (AMH) levels | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the endocrine marker of ovarian reserve
Change of Inhibin B levels | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the endocrine marker of ovarian reserve
Change of antral follicular count (AFC) | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the US marker of ovarian reserve

SECONDARY OUTCOMES:
Change of CA -125 levels | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the inflammatory marker
Change of interleukin-6 (IL-6) levels | 2nd to 5th day of the cycle in which laparoscopy is performed and 2nd to 5th day of the cycle in 6th month after laparoscopy
  as the inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana S Spremovic-Radjenovic, Professor, Principal Investigator — CCSerbia, School of Medicine, University of Belgrade
Locations (3):
- Serbia (3):
  - General Hospital of Subotica, Subotica, Vojvodina
  - CCSerbia, Clinic for Gynecology and Obstetrics, School of Medicine, University of Belgrade, Belgrade
  - Department of Laboratory Medicine ''Konzilijum'', Belgrade

REFERENCES:
- [Background] Jadoul P, Kitajima M, Donnez O, Squifflet J, Donnez J. Surgical treatment of ovarian endometriomas: state of the art? Fertil Steril. 2012 Sep;98(3):556-63. doi: 10.1016/j.fertnstert.2012.06.023. Epub 2012 Jul 3. PMID 22763094
- [Background] Kitajima M, Defrere S, Dolmans MM, Colette S, Squifflet J, Van Langendonckt A, Donnez J. Endometriomas as a possible cause of reduced ovarian reserve in women with endometriosis. Fertil Steril. 2011 Sep;96(3):685-91. doi: 10.1016/j.fertnstert.2011.06.064. Epub 2011 Jul 29. PMID 21802672
- [Background] Muzii L, Di Tucci C, Di Feliciantonio M, Marchetti C, Perniola G, Panici PB. The effect of surgery for endometrioma on ovarian reserve evaluated by antral follicle count: a systematic review and meta-analysis. Hum Reprod. 2014 Oct 10;29(10):2190-8. doi: 10.1093/humrep/deu199. Epub 2014 Aug 1. PMID 25085800
- [Background] Raffi F, Metwally M, Amer S. The impact of excision of ovarian endometrioma on ovarian reserve: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2012 Sep;97(9):3146-54. doi: 10.1210/jc.2012-1558. Epub 2012 Jun 20. PMID 22723324
- [Background] Somigliana E, Berlanda N, Benaglia L, Vigano P, Vercellini P, Fedele L. Surgical excision of endometriomas and ovarian reserve: a systematic review on serum antimullerian hormone level modifications. Fertil Steril. 2012 Dec;98(6):1531-8. doi: 10.1016/j.fertnstert.2012.08.009. Epub 2012 Sep 10. PMID 22975114
- [Background] Hart RJ, Hickey M, Maouris P, Buckett W. Excisional surgery versus ablative surgery for ovarian endometriomata. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004992. doi: 10.1002/14651858.CD004992.pub3. PMID 18425908